CLINICAL TRIAL: NCT00896545
Title: Development of an Early Intervention for the Prevention of Childhood Obesity
Brief Title: Early Childhood Prevention of Childhood Overweight
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: William Stewart Agras, Principal Investigator, Stanford University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SU-04072009-2158
Record Dates: First submitted 2009-05-07; First posted 2009-05-11 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 5-keys feeding program (Experimental): Counseling in small groups aimed at enhancing children's self control over eating
  Interventions: Behavioral: 5-keys counseling; Behavioral: Lifestyle counseling
- Healthy lifestyle counseling (Active Comparator): Counseling in small groups aimed at achieving healthy eating patterns aimed at both the family and young children
  Interventions: Behavioral: Lifestyle counseling

INTERVENTIONS:
Behavioral: 5-keys counseling — 5-session small group intervention
  Arms: 5-keys feeding program
Behavioral: Lifestyle counseling — 5-session small group behavioral intervention

SUMMARY:
You are invited to participate in a research study to understand more about childhood obesity and how to prevent it. We hope to learn how families influence each others eating habits.

DETAILED DESCRIPTION:
This study aims to understand more about childhood obesity and how to prevent it. Two different methods of prevention will be tested and participants will be allocated at random to one of these methods. The investigators hope to learn how families influence each others eating habits.

Participants in this study will attend a series of five classes, once a week for five weeks, on the topic of child feeding. The aim of the classes is to learn how to feed your child so as to prevent future eating and weight problems. The research component includes filling out some surveys before classes begin and at the end of the last class. Classes are small and interactive so that parents have a chance to voice concerns and get feedback.

ELIGIBILITY:
Inclusion Criteria:

* One or both parents with BMI > or = to 27.5
* Healthy child ages 2-4 years

Exclusion criteria.

- Inadequate understanding of the English language

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2008-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Parental control of feeding | 5-weeks
  Assessed by Questionnaire pre and post treatment.

SECONDARY OUTCOMES:
Daily patterns of child and family meals | 1-week
  Assessed by questionnaire pre and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: William Stewart Agras, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States